CLINICAL TRIAL: NCT06348940
Title: Effects of Behavioral Activation on Negative Emotions, Cancer-related Symptoms and Clinical Indicators in Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Huaidong Cheng, Professor, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 83242392
Record Dates: First submitted 2024-03-23; First posted 2024-04-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cancer Patients

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral activation + Care as usual (Experimental): Cohort 1-5: Intervention Group
  Interventions: Behavioral: behavioral activation
- Care as usual (No Intervention): Cohort 1-5: Control Group

INTERVENTIONS:
Behavioral: behavioral activation — Behavioral activation, an emerging psychological intervention approach, has potential in alleviating negative emotions among cancer patients. The intervention group underwent an eight-week behavioral activation program designed to promote engagement in meaningful activities that are physically and emotionally rewarding while reducing involvement in maladaptive emotional cycles.
  Arms: Behavioral activation + Care as usual

SUMMARY:
The majority of cancer patients experience varying degrees of psychological distress and physical symptoms due to the presence of cancer or the process of treatment. These symptoms are closely associated with inflammatory markers and patient prognosis, highlighting the urgent need for effective psychological intervention methods. Behavioral activation, an emerging psychological intervention approach, requires further investigation regarding its potential in alleviating negative emotions among cancer patients. Therefore, the objective of this study is to investigate whether (1) behavioral activation can ameliorate negative emotions and physical symptoms in cancer patients; (2) behavioral activation can contribute to improved survival outcomes for these patients; and (3) behavioral activation can enhance NLR levels and other clinical indicators among individuals with cancer.

The investigators aimed to recruit esophageal and gastric cancer, colorectal cancer, and non-small cell lung cancer (NSCLC) patients. These patients were recruited from the Department of Oncology at the Second Affiliated Hospital of Anhui Medical University between March 2023 and November 2023. They are divided into seven cohorts. Cohorts 1-5 are randomized control trials and within each cohort, patients were randomly allocated into two groups: an intervention group (behavioral activation+care as usual, BA+CAU) and a control group (care as usual, CAU). The intervention group underwent an eight-week behavioral activation program (see Detailed Description) designed to promote engagement in meaningful activities that are physically and emotionally rewarding while reducing involvement in maladaptive emotional cycles. Both the intervention group and the control group received standard care along with conventional treatment for their respective cancers. Cohorts 6-7 are prospective cohort studies, in addition to the aforementioned groups, and include an additional control group. Detailed information for each cohort is provided in Detailed Description.

This study aims to demonstrate the significant efficacy of behavioral activation in improving negative emotions, somatic symptoms, quality of life, and clinical inflammatory indicators among cancer patients. Furthermore, it may potentially enhance patient survival rates, thereby offering a novel approach for psychological intervention in cancer patients and contributing to multidisciplinary treatment and management strategies. The intervention measures employed in this study do not involve any pharmacological treatments or hazardous activities. For illiterate or less educated patients, the informed consent process and questionnaire collection will be conducted using methods that ensure their full comprehension (e.g., verbal explanations, visual aids). Additionally, patients with evident cognitive impairments were excluded from the study.

The investigators have implemented a questionnaire system on the WJX website (https://www.wjx.cn/) to collect patient information through both paper and electronic questionnaires. The psychological measurement questionnaires are stored electronically, while socio-demographic data and clinical indicators are collected in the hospital's medical record management system. Subsequently, all data is summarized and saved in local Excel files and SPSS files for specialized analysis by data analysts. Patient names are anonymized within the database, ensuring strict confidentiality of personal information such as contact details and home address.

Possible statistical methods include descriptive statistical analysis, generalized estimating equation or repeated measures analysis of variance, structural equation modeling, correlation analysis and regression, survival analysis, etc.

DETAILED DESCRIPTION:
Study cohort:

Cohort 1: A randomized controlled trial was conducted to investigate the potential of BA in mitigating stigma among patients with advanced esophageal and gastric cancer, while also enhancing their quality of life. (Primary measure: Stigma, Secondary measure: Quality of life)

Cohort 2: A randomized controlled trial was conducted to investigate the potential of BA in mitigating psychological distress among patients with all stages of esophageal and gastric cancer and the mediating role of self-efficacy. (Primary measure: Psychological distress, Secondary measure: Anxiety symptoms, Self-efficacy, Effects of BA)

Cohort 3: A randomized controlled trial was conducted to investigate the potential of BA in mitigating depression symptoms among patients with colorectal cancer and the mediating role of physical activity. (Primary measure: Depression symptoms, Physical activity, Secondary measure: Quality of life, Psychological distress, Anxiety symptoms, Effects of BA)

Cohort 4: A randomized controlled trial was conducted to investigate the potential of BA in mitigating cancer-related fatigue among patients with non-small cell lung cancer (NSCLC). (Primary measure: Cancer-related fatigue, Secondary measure: Quality of life, Psychological distress, Depression symptoms, Anxiety symptoms, Effects of BA)

Cohort 5: A randomized controlled trial was conducted to investigate the potential of BA in mitigating fear of cancer recurrence among patients with non-small cell lung cancer (NSCLC). (Primary measure: Fear of cancer recurrence, Secondary measure: Quality of life, Psychological distress, Depression symptoms, Anxiety symptoms, Social Support, Self-efficacy)

Cohort 6: A prospective cohort study was conducted to investigate the potential of BA in alleviating emotional distress, reducing inflammation markers, and improving outcomes in patients with advanced digestive system cancers (esophageal cancer, gastric cancer, and colorectal cancer) receiving first-line Immune Checkpoint Inhibitors (ICIs) therapy through the categorization into three groups: those experiencing pre-treatment emotional distress without BA intervention, those experiencing pre-treatment emotional distress with BA intervention, and those without pre-treatment emotional distress without BA intervention. (Primary measure: Progression-Free Survival, PFS)

Cohort 7: A prospective cohort study was conducted to investigate the potential of BA in alleviating emotional distress, reducing inflammation markers, and improving outcomes in patients with non-small cell lung cancer (NSCLC) receiving first-line Immune Checkpoint Inhibitors (ICIs) therapy through the categorization into three groups: those experiencing pre-treatment emotional distress without BA intervention, those experiencing pre-treatment emotional distress with BA intervention, and those without pre-treatment emotional distress without BA intervention. (Primary measure: Progression-Free Survival, PFS)

Study procedure:

This study was evaluated by experts in the field, including two psychologists and one oncologist to ensure its scientificity and feasibility. The BA intervention was administered 8 times, once a week. Each session lasted for 15-30 min. All the interventions were conducted by the same psychological consultant. The first BA intervention for each patient was conducted in person, with a psychological consultant in a separate treatment room. Thereafter, the psychological intervention sessions for most patients were conducted via audio calls or video conferencing means (WeChat or phone). With informed consent from all participants, each audio call was recorded, and these recordings served as the basis for the examiner's assessment of the quality of the intervention. If the BA intervention could not be conducted at the scheduled time due to patients' physical condition or other reasons, it was rescheduled within 3 to 5 days from the specified intervention time. In addition to the BA intervention, the BA+CAU group received comparable cancer care and treatment to that of the control group.

The aim of BA is to promote engagement in meaningful and pleasurable activities while reducing those that perpetuate negative emotional cycles. The investigators developed a 8-week program based on the Brief Behavioral Activation Treatment for Depression: Revised Treatment Manual. Patients were assessed weekly and instructed to keep track of their activities from the past week, rating each activity for its level of pleasure and meaning, as well as providing an overall rating for the week. Based on these scores, patients can identify which activities are beneficial or detrimental to their mental health and create a plan to increase positive activities in the following week. If they encounter difficulties achieving these goals, the investigators encourage them to break down larger objectives into smaller specific tasks or make "contracts" with others for support. Additionally, if patients are less active, the investigators suggest selecting some activities from our list (family, social, religious, etc.) as targets.

8-week program

Sessions Key elements Weekly Assignments Session1 (Special session) Offline intervention 1.Discussion of Depression 2.Introduction to Treatment Rationale. What about stressful life events and loss in participant's life? 3.Introduction to Daily Monitoring: (1) Importance and enjoyment (or meaning and happiness) ratings. (2) When should participants complete the Daily Monitoring Form? 4.Important Points About the Structure of This Treatment Complete Daily Monitoring Form Session 2 (Special session) Via telephone or Wechat: 1.Daily Monitoring: Review Assignment, Troubleshooting 2.Treatment Rationale: Review 3.Complete Life Areas, Values, Activities Inventory (Appendix) 1. Complete Daily Monitoring 2. Review and edit Life Areas, Values, and Activities Inventory Session 3 (Special session) Via telephone or Wechat: 1.Daily Monitoring: Review Assignment 2.Life Areas, Values, and Activities Inventory: Review assignment 3.Activity Selection and Ranking 1.Daily monitoring 2.Continue to review and edit Life Areas, Values, and Activities Inventory 3. Review and edit activity selection and ranking Session 4 (Special session) Via telephone or Wechat: 1.Daily Monitoring: Review Assignment 2.Daily Monitoring with Activity Planning Daily Monitoring with activity planning for upcoming week Session 5 (Special session) Via telephone or Wechat: 1.Daily Monitoring With Activity Planning: Review Assignment 2.Contract: Ensure the timely completion of activities through effective collaboration with other people 3.Daily Monitoring With Activity Planning for the Upcoming Week 1.Daily monitoring with activity planning for the upcoming week 2.Continue adding/editing contracts Session 6 (Maintenance Session) Via telephone or Wechat: 1.Daily Monitoring With Activity Planning: Review Assignment 2.Life Areas, Values, and Activities Inventory: Concept Review and Edit 3.Daily Monitoring With Activity Planning for the Upcoming Week 1.Daily monitoring with activity planning for the upcoming week 2.Continue adding/editing Contracts Session 7 (Maintenance Session) Via telephone or Wechat: 1.Daily Monitoring With Activity Planning: Review Assignment 2.Life Areas, Values, and Activities Inventory: Concept Review and Edit 3.Daily Monitoring With Activity Planning for the Upcoming Week 1.Daily monitoring with activity planning for the upcoming week 2.Continue adding/editing contracts Session 8 (Maintenance Session) Via telephone or Wechat: 1.Daily Monitoring With Activity Planning: Review Assignment 2.Daily Monitoring With Activity Planning for the Upcoming Week 3.Preparing for the End of Treatment 1.Daily monitoring with activity planning for the upcoming week 2.Continue adding/editing contracts

ELIGIBILITY:
Cohort 1:

Inclusion criteria:

(Patients who)

* Had to meet the diagnostic criteria for esophageal or gastric cancer through clinical, pathological, and imaging examinations,
* Should have no history of prior psychological intervention,
* Karnofsky Performance Status (KPS) score should be equal to or greater than 80 points,
* Were required to complete the questionnaire independently or with assistance from others if needed,
* Were consistently admitted to the hospital for tumor treatment, with an average time interval of approximately one month between each hospitalization,
* Were reporting stigma and its possible causes, the average score of the Social Impact Scale exceeded 1,
* Were of legal age, 18 years or older.

Exclusion criteria:

(Patients who)

* With severe intellectual disabilities or other communication difficulties that hindered normal interaction,
* With an expected survival time of less than 4 months,
* Were Cachexia or severely debilitated,
* With fractures, serious heart dysfunction, or significant comorbidities involving the liver, kidneys, and other organs/tissues,
* With early esophageal or gastric cancer (tumor tissue has not infiltrated the muscularis propria layer),
* With a history of using psychotropic or psychoactive drugs.

Cohort 2:

Inclusion criteria:

(Patients who)

* Had to meet the diagnostic criteria for esophageal or gastric cancer through clinical, pathological, and imaging examinations,
* Should have no history of prior psychological intervention,
* Karnofsky Performance Status (KPS) score should be equal to or greater than 80 points,
* Were required to complete the questionnaire independently or with assistance from others if needed,
* Were consistently admitted to the hospital for tumor treatment, with an average time interval of approximately one month between each hospitalization,
* Psychological Distress Thermometer (DT) score should be equal to or greater than 4 points,
* Were of legal age, 18 years or older.

Exclusion criteria:

(Patients who)

* With severe intellectual disabilities or other communication difficulties that hindered normal interaction,
* With an expected survival time of less than 4 months,
* Were Cachexia or severely debilitated,
* With fractures, serious heart dysfunction, or other severe medical conditions,
* With a history of using psychotropic or psychoactive drugs.

Cohort 3:

Inclusion criteria:

* Age ≥18 years with sufficient hearing and vision capabilities,
* Good activity ability, KPS score ≥80,
* No history of psychological intervention,
* Clear diagnosis of colorectal cancer with an expected survival of ≥6 months,
* Hospital Anxiety and Depression Scale (HADS) depression score ≥8,
* Sufficient ability to record and communicate independently or with family help,
* Regular hospital visits for treatment or examination.

Exclusion Criteria:

* Known neurological diseases affecting cognition,
* Previous use of medication to improve cognitive function,
* Combined with other severe chronic diseases or organ damage.

Termination Criteria:

* Severe adverse events or reactions making it difficult to continue intervention,
* Physical or mental symptoms worsen, or new symptoms emerge, making it impossible to continue intervention,
* The patient wishes to stop the intervention,
* More than three weeks between sessions,
* Use of psychotropic drugs at the discretion of the attending physician during the intervention or waiting period,
* Meeting exclusion criteria during the waiting period,
* Other reasons deemed necessary by the attending physician to stop the intervention.

Cohort 4:

Inclusion criteria:

* Diagnosis of primary non-small cell lung cancer confirmed through clinical, pathological, and imaging examinations, and awareness of their condition;
* Absence of prior psychological interventions;
* PFS score of ≥1;
* Age of 18 years or older at the time of diagnosis and possessing adequate audiovisual capabilities to complete the questionnaire and intervention procedures.

Exclusion criteria:

* Individuals with severe intellectual disabilities or communication impairments;
* Patients with an estimated survival time of less than 4 months;
* Patients with fractures, severe cardiac insufficiency, or other serious medical conditions.

Termination criteria:

* Occurrence of serious adverse events or reactions hindering intervention continuation;
* Patient's expressed desire to discontinue the intervention;
* Inter-meeting intervals of at least three weeks;
* Regular usage of fatigue or psychotropic medications as deemed appropriate by the attending physician during program implementation or the waiting period;
* Compliance with exclusion criteria during the waiting period;
* Any other reasons determined necessary by the attending physician to cease the intervention.

Cohort 5:

Inclusion criteria:

* Meet the diagnostic criteria for primary NSCLC through clinical, pathological, and imaging examinations and are aware of their diagnosis;
* Have not received any prior psychological intervention;
* Have a FCRI-SF score of ≥13 points;
* Are 18 years of age or older at the time of diagnosis and have sufficient auditory and visual abilities to complete the questionnaire tests and intervention procedures.

Exclusion criteria:

* Individuals with severe cognitive impairments or other communication difficulties;
* Patients with an estimated survival time of less than 4 months;
* Patients with fractures, severe cardiac insufficiency, or other serious comorbidities.

Termination criteria:

* Serious adverse events or adverse reactions that make it difficult to continue the intervention;
* Patient requests to discontinue the intervention;
* At least three weeks elapsing between sessions;
* Regular use of fatigue or psychotropic medications, as determined by the attending physician, during the implementation of the program or during the waiting period;
* Meeting the exclusion criteria during the waiting period;
* Other reasons deemed necessary by the attending physician to discontinue the intervention.

Cohort 6:

Inclusion criteria:

* Meet the diagnostic criteria for digestive system cancers (esophageal cancer, gastric cancer, or colorectal cancer) through clinical, pathological, and imaging examinations;
* Karnofsky Performance Status (KPS) score should be equal to or greater than 80 points;
* Systematic treatments naive ( e. g., chemotherapy, anti-angiogenic drugs, targeted drugs, and immunotherapy);
* Presence of at least one measurable lesion according to the Response Evaluation Criteria in Advanced Solid Tumors version 1.1 (RECIST v1.1);
* Receiving PD-1/PD-L1 inhibitors monotherapy or combination with chemotherapy;
* Informed and agreed to participate in the study;
* Required to complete the questionnaire independently or with assistance from others if needed;
* Legal age, 18 years or older.

Exclusion criteria:

* Oncogene-driver positive;
* Resectable early esophageal or gastric cancer (tumor tissue has not infiltrated the muscularis propria layer);
* Combined with other malignant tumors in the past 3 years;
* Concurrent acute or chronic psychiatric disorders;
* Current receiving anti-depressive or anti-anxiety therapy or other psychotropic drugs;
* Previous treatment with other clinical drug trials;
* Patients with symptomatic brain metastasis;
* Severe intellectual disabilities or other communication difficulties that hindered normal interaction.

Termination criteria:

* Serious adverse events or adverse reactions that make it difficult to continue the intervention;
* Patient requests to discontinue the intervention;
* Regular use of psychotropic or psychoactive drugs, as determined by the attending physician, during the implementation of the program or during the waiting period;
* Other reasons deemed necessary by the attending physician to discontinue the intervention.

Cohort 7:

Inclusion criteria:

* Meet the diagnostic criteria for NSCLC through clinical, pathological, and imaging examinations;
* Karnofsky Performance Status (KPS) score should be equal to or greater than 80 points;
* Unresectable locally advanced, metastatic, or recurrent stage ⅢB-Ⅳ based on AJCC TNM staging 8th edition;
* Systematic treatments naive ( e. g., chemotherapy, anti-angiogenic drugs, targeted drugs, and immunotherapy);
* Presence of at least one measurable lesion according to the Response Evaluation Criteria in Advanced Solid Tumors version 1.1 (RECIST v1.1);
* Receiving PD-1/PD-L1 inhibitors monotherapy or combination with chemotherapy;
* Informed and agreed to participate in the study;
* Required to complete the questionnaire independently or with assistance from others if needed;
* Legal age, 18 years or older.

Exclusion criteria:

* Oncogene-driver positive;
* Combined with other malignant tumors in the past 3 years;
* Concurrent acute or chronic psychiatric disorders;
* Current receiving anti-depressive or anti-anxiety therapy or other psychotropic drugs;
* Previous treatment with other clinical drug trials;
* Patients with symptomatic brain metastasis;
* Severe intellectual disabilities or other communication difficulties that hindered normal interaction.

Termination criteria:

* Serious adverse events or adverse reactions that make it difficult to continue the intervention;
* Patient requests to discontinue the intervention;
* Regular use of psychotropic or psychoactive drugs, as determined by the attending physician, during the implementation of the program or during the waiting period;
* Other reasons deemed necessary by the attending physician to discontinue the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic data | Day 0
  The sociodemographic data includes gender, age, smoking, drinking, working, marital status, and education level. This information is extracted from the medical record.
Status of Tumor | Day 0
  The status of tumor encompasses the primary tumor site, TNM stage-based tumor staging, histological subtype of the tumor, as well as the past, present, and future treatment strategies for the neoplasm. This information is extracted from the medical record.
Body Mass Index, BMI | Day 0, Month 1, Month 2, Month 6 and Month 12
  The Body Mass Index (BMI) is a widely accepted international standard for assessing adiposity and overall health status in individuals. It is calculated by dividing an individual's weight by the square of their height, expressed in kilograms per square meter (kg/m^2). This information is extracted from the medical record.
Biochemical index | Day 0, Month 1, Month 2, Month 6 and Month 12
  Biochemical index includes blood glucose, triglyceride and total cholesterol, which reflect the metabolic level in the body, expressed in mmol/L. This information is extracted from the medical record. This information is extracted from the medical record.
Blood Pressure, BP | Day 0, Month 1, Month 2, Month 6 and Month 12
  The measurement of blood pressure is typically presented as the ratio between systolic and diastolic pressures, expressed in millimeters of mercury (mmHg). This information is extracted from the medical record.
Nutritional Risk Screening, NRS | Day 0, Month 1, Month 2, Month 6 and Month 12
  NRS is a recommended method by the European Society for Parenteral and Enteral Nutrition to assess nutritional risk in hospitalized patients, consisting of three components: nutritional status, disease severity, and age. The total score ranges from 0-7 points with higher scores indicating poorer nutritional status. A total score ≥3 points indicates the presence of nutritional risk requiring nutritional support while a total score <3 points necessitates weekly review of the patient's nutritional assessment; if subsequent reviews yield a score ≥3 points, then initiation of the nutritional support program is warranted.
Visual Analogue Scale, VAS | Day 0, Month 1, Month 2, Month 6 and Month 12
  VAS is a widely utilized tool for pain assessment in clinical practice in China. This method involves employing a 10cm long sliding ruler, featuring 10 gradations on one side and "0" and "10" at the opposing ends. A score of 0 indicates the absence of pain, while a score of 10 represents the utmost intolerable pain.
Karnofsky Performance Status Scale, KPS | Day 0, Month 1, Month 2, Month 6 and Month 12
  KPS is utilized for the evaluation of cancer patients' physical condition and daily functional capacity. The total score ranges from 0 to 100, with higher scores indicating improved overall health, enhanced physical abilities, better tolerance towards treatment-related side effects, and consequently a greater potential for comprehensive therapeutic interventions.
Psychological Distress Thermometer (DT) | Day 0, Month 1, Month 2, Month 6 and Month 12
  Psychological distress is assessed using the DT. The DT is a self-assessment of the level of psychological distress experienced in the past week (including the day of filling in this questionnaire). It covers practical, family, emotional, spiritual/religious and physical problems. The scale ranges from 0 to 10. The higher the score, the greater the level of psychological distress or psychological distress.
Hospital anxiety and depression scale (HADS) | Day 0, Month 1, Month 2, Month 6 and Month 12
  Anxiety and depression were assessed using the HADS. The HADS scale is mainly used for screening anxiety and depression in general hospital patients. It includes two subscales, HADS-A and HADS-D, with a total of 14 items, including 7 items for anxiety (A) and 7 items for depression (D). Each item is scored on a 4-level scale according to the frequency of symptoms in the past month. Each item has a total of four levels, ranging from 0 to 3, with higher scores indicating more severe anxiety or depression symptoms. The total scores for anxiety and depression are 0-21.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Day 0, Month 1, Month 2, Month 6 and Month 12
  Quality of life was assessed using the EORTC QLQ-C30. The EORTC QLQ-C30 is a cancer-specific tool that contains 30 items. The EORTC QLQ-C30 includes five important functional areas -- physical, emotional, role, cognitive, and social; two items assess global quality of life; three symptom scales assess fatigue, vomiting, and pain; and six subscales to assess dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial difficulties. Higher scores on the functional scales represent higher levels of functioning, meaning healthier cancer patients, while higher scores on the symptom scales or items represent higher levels of symptoms or problems, or less healthy cancer patients.
Pittsburgh sleep quality index (PSQI) | Day 0, Month 1, Month 2, Month 6 and Month 12
  The Pittsburgh Sleep Quality Index (PSQI) is used to assess subjective sleep quality over the past month. The PSQI consists of 19 self-rated items and 7 dimensions: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, hypnosis use, and daytime dysfunction. The scores range from 0 to 3 and the total score is 0 to 21; higher scores indicate poorer sleep quality.
Revised Piper Fatigue Scale (PFS-R) | Day 0, Month 1, Month 2, Month 6 and Month 12
  Cancer-related fatigue was assessed using the PFS-R. The scale consists of 22 items and 5 open-ended questions, and patients were evaluated using a scale of 0 to 10, with the final score as total score/item number. The PFS-R described four dimensions of subjective fatigue according to the following subscales: behavioral severity subscale (6 items), cognitive severity subscale, emotional meaning subscale (5 items), and sensory/emotional severity subscale (5 items). Fatigue was divided into three grades according to the score: mild fatigue (1-3 points), moderate fatigue symptoms (4-6 points), and severe fatigue symptoms (7-10 points).
International physical activity questionnaire (IPAQ) | Day 0, Month 1, Month 2, Month 6 and Month 12
  The physical activity level was assessed by the short version of the International Physical Activity Questionnaire (IPAQ). There were seven questions in total, six of which asked about the physical activity of individuals. The question structure was the same as that of the long version of the IPQ, except for the activity intensity part. The short version of the IPQ was divided into walking, moderate intensity and high intensity to ask about the weekly frequency and cumulative time of activities of different intensity, taking into account the four physical activity levels of work, transportation, housework and gardening, and leisure. Participants were categorized into low, moderate, and high physical activity groups based on their overall level of physical activity as well as the frequency and duration of daily physical activities over a span of one week.
Brief Resilient Coping Scale (BRCS) | Day 0, Month 1, Month 2, Month 6 and Month 12
  The Brief Resilient Coping Scale was used to assess resilience. It has four items and uses a 5-point Likert scale "from '1' = does not describe me at all to '5' = describes me very much."25 The total score ranges from 4 to 20; higher scores indicate greater resilience.
Multidimensional Scale of Perceived Social Support (MSPSS) | Day 0, Month 1, Month 2, Month 6 and Month 12
  Social support was assessed using the Perceived Social Support Multidimensional Scale. The scale includes 12 self-rated items and uses a 7-point scoring method, with scores ranging from strongly disagree to strongly agree, with higher scores indicating higher perceived social support. This study used the scale to assess the perceived degree of support from family, friends and others.
General Self-Efficacy Scale (GSES) | Day 0, Month 1, Month 2, Month 6 and Month 12
  Self-efficacy was assessed using the General Self-Efficacy Scale. The scale consists of 10 items, each of which is scored between 1 and 4, and the total score is 10-40 divided by 10. The higher the score, the higher the self-efficacy.
The activation subscale of Behavioral Activation for Depression Scale (BADS-A) | Day 0, Month 1, Month 2, Month 6 and Month 12
  The effectiveness of the BA intervention was assessed using the BADS-A, a 7-item scale that allows each item to be scored on a scale of 0 to 6 (from "none at all" to "completely"), with a total score of 0 to 42. The higher the score, the better the BA intervention.
Social Impact Scale (SIS) | Day 0, Month 1, Month 2, Month 6 and Month 12
  The Social Impact Scale is used to evaluate the stigma of patients with chronic diseases such as cancer. The scale has 24 items, including 4 dimensions, which are social exclusion, economic discrimination, internal stigma and social isolation. The scale adopts the Likert 4-point scoring method, with 1-4 points from "strongly disagree" to "strongly agree", and the total score ranges from 24 to 96. The higher the score, the greater the stigma of patients.
Fear of Cancer Recurrence Inventory- Short Form (FCRI-SF) | Day 0, Month 1, Month 2, Month 6 and Month 12
  Fear of recurrence was assessed with the Fear of Cancer Recurrence Inventory- Short Form, which consists of 9 questions and is graded on a 0 to 4 scale with a total score of 0 to 36, with higher scores indicating greater fear of recurrence, with a cutoff score of 13 for high-level FCR.
The Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog) | Day 0, Month 1, Month 2, Month 6 and Month 12
  The FACT-Cog is used to assess perceived cognitive function and its impact on quality of life in cancer patients. It includes 37 items across four dimensions (subjective cognitive impairment, evaluation by others, subjective cognitive ability, and impact of cognitive impairment on quality of life), with each item scored on a scale of 0 to 5, ranging from never/not at all (0) to several times/very often (4). The total score is 0 to 148, with lower scores indicating greater cognitive impairment.
Time of Progression-free survival (PFS) | 1 year
  Progression-free survival (PFS) is the time from randomization to the first progression or death from any cause. The criteria for tumor progression are based on the RECIST 1.1 version.
Time of Time to progression (TTP) | 1 year
  Time to progression (TTP) is the time from randomization to any aspect of tumor progression. The criteria for tumor progression are based on the RECIST 1.1 version.
Objective Response Rate (ORR) | 1 year
  The proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Concentration of C-reactive protein (CRP) | 1 year
  C-reactive protein (CRP) expressed in mg/L, serves as a non-specific inflammatory biomarker with higher values indicating elevated levels of systemic inflammation. This information is extracted from the medical record.
Value of Neutrophils to lymphocytes ratio (NLR) | 1 year
  NLR is an inflammatory marker, which is the ratio of neutrophils to lymphocytes. The higher the value is, the higher the inflammatory level may be. This information is extracted from the medical record.
Value of Platelet-lymphocyte ratio (PLR) | 1 year
  PLR is an inflammatory marker, a ratio of platelets to lymphocytes. A higher value of it indicates a higher level of inflammation in the body. This information is extracted from the medical record.
Value of Monocyte-lymphocyte ratio (MLR) | 1 year
  MLR is an inflammatory indicator, which is the ratio of macrophages and lymphocytes. The higher the value is, the higher the inflammatory level in the body is. This information is extracted from the medical record.
Value of Systemic immune inflammation index (SII) | 1 year
  SII is an inflammatory indicator, which is calculated as follows: SII=(neutrophil×platelet)/lymphocytes. A higher value indicates an elevated level of inflammation within the body. This information is extracted from the medical record.
Value of Pan-immune inflammation value (PIV) | 1 year
  PIV is an inflammatory indicator, which is equal to neutrophils × monocytes × platelets/lymphocytes. The higher the value is, the higher the inflammatory level in the body is. This information is extracted from the medical record.
Value of eosinophil fraction | 1 year
  The eosinophil fraction is a potential inflammation and tumor prognostic indicator, which equals the ratio of eosinophil absolute value to the total white blood cell count. The higher the value of this fraction, the better the tumor prognosis may be. The information has been extracted from the medical record and evaluated longitudinally.
Value of prognostic nutritional index (PNI) | 1 year
  PNI is a potential inflammation and tumor prognostic indicator, which is equal to albumin level (g/L) + 5 × absolute value of lymphocyte counts. The higher the value of this index, the better the tumor prognosis may be. The information has been extracted from the medical record and evaluated longitudinally.
Value of the modified Glasgow prognostic score (mGPS) | 1 year
  mGPS is a potential inflammation and tumor prognostic indicator, which based on serum C-reactive protein (CRP) and albumin. Patients were assigned mGPS = 0 if normal serum C-reactive protein (CRP, ≤10 mg/L) and albumin levels (≥35 g/L) were observed. Patients were assigned mGPS = 1 if elevated CRP without hypoalbuminemia (CRP > 10 mg/L and albumin ≥35 g/L) was diagnosed. If CRP >10 mg/L and albumin <35 g/L, mGPS = 2. The higher the score, the worse the tumor prognosis may be. The information has been extracted from the medical record and evaluated longitudinally.
Concentration of Carcinoembryonic antigen (CEA) | 1 year
  Carcinoembryonic antigen (CEA) is a broad-spectrum tumor marker, commonly found in gastrointestinal tumors as well as breast and lung cancers. Normal values are generally <5.0ng/ml. This information is extracted from the medical record.
Concentration of Carbohydrate antigen 19-9 (CA19-9) | 1 year
  Carbohydrate antigen 19-9 (CA19-9) is a tumor marker associated with pancreatic, gallbladder, colon, and stomach cancers, with a normal value of <37kU/L. This information is extracted from the medical record.
Concentration of Carbohydrate antigen 72-4 (CA72-4) | 1 year
  Carbohydrate antigen 72-4 (CA72-4) is one of the tumor markers for the detection of gastric cancer and various digestive tract cancers. The detection of gastric cancer exhibits a high level of specificity, with a cut-off value set at >6 U/mL. This information is extracted from the medical record.
Concentration of Neuron-specific enolase (NSE) | 1 year
  Neuron-specific enolase (NSE) is a specific marker for tumors such as small cell lung cancer (SCLC), with normal value <16.3ng/ml. This information is extracted from the medical record.
Concentration of Squamous cell carcinoma associated antigen (SCC) | 1 year
  Squamous cell carcinoma associated antigen (SCC) is a tumor marker associated with squamous cell carcinomas such as lung squamous cell carcinoma and esophageal squamous cell carcinoma, with a cut-off value of 2.5μg/L. This information is extracted from the medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li A, Huang R, Ge H, Liu D, Liu S, Jia Y, Chai J, Zheng X, Liu L, Gan C, Xu J, Cheng L, Zhang M, Cheng H. Exploring the impact and mechanisms of behavioral activation on sleep disorders in colorectal cancer: a randomized controlled trial. J Cancer Res Clin Oncol. 2024 Dec 20;151(1):12. doi: 10.1007/s00432-024-06065-x. PMID 39706981
- [Derived] Huang R, Ge H, Nie G, Li A, Liu L, Cheng L, Zhang M, Cheng H. Effect of Behavioral Activation on Stigma and Quality of Life in Patients With Advanced Esophageal and Gastric Cancer: A Randomized Controlled Trial. Psychooncology. 2024 Nov;33(11):e70021. doi: 10.1002/pon.70021. PMID 39547955
- [Derived] Huang R, Li A, Ge H, Liu L, Cheng L, Zhang M, Cheng H. Impacts and Pathways of Behavioral Activation on Psychological Distress Among Patients Diagnosed With Esophageal and Gastric Cancer in China: A Randomized Controlled Trial. Cancer Med. 2024 Oct;13(19):e70314. doi: 10.1002/cam4.70314. PMID 39404168